CLINICAL TRIAL: NCT06927492
Title: Effects of Cognitive Sensorimotor Training With Whole Body Vibration on Cognition and Balance in Older Adults With Cognitive Impairment
Brief Title: Cognitive Sensorimotor Training With Whole Body Vibration for Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0260 Tooba Saher
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Impairment
Keywords: Sensory motor training; WBV; Functional mobility; Short performance battery
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Cognitive Sensorimotor training along with whole body vibration (Experimental): This group will receive sensorimotor training with cognitive dual-task training in addition to whole body vibration. The participants will perform 36 sessions (3 times per week on alternate days over 12 weeks). The duration of one session for each group will be 60 minutes,
  Interventions: Other: Cognitive Sensorimotor training along with whole body vibration
- B: Cognitive Sensorimotor training (Experimental): This group will receive sensorimotor training with cognitive dual task training simultaneously. The participants will perform 36 sessions (3 times per week on alternate days over 12 weeks). The duration of one session for each group will be 60 minutes,
  Interventions: Other: Cognitive Sensorimotor training

INTERVENTIONS:
Other: Cognitive Sensorimotor training along with whole body vibration — This group will receive sensorimotor training with cognitive dual-task training in addition to whole body vibration. The participants will perform 36 sessions (3 times per week on alternate days over 12 weeks). The duration of one session for each group will be 60 minutes, The whole-body vibration will be administered using a vibration machine. This includes asking the patient to stand barefoot on the vibrator platform evenly distributing their body weight on both feet with knees bent at 20 degrees as flexing of knees is a common postural adaptation used to minimize transmission of vibration to the head. The patients will receive the whole body vibration at 30Hz consisting of three sessions per week with at least one day between sessions for 12 weeks. The time for each session will be 15 minutes (five bouts of 2 min) . There will be a rest of 1 minute between each bout of vibration therapy.
  Arms: A: Cognitive Sensorimotor training along with whole body vibration
Other: Cognitive Sensorimotor training — This group will receive sensorimotor training with cognitive dual task training simultaneously. The participants will perform 36 sessions (3 times per week on alternate days over 12 weeks). The duration of one session for each group will be 60 minutes,
  Arms: B: Cognitive Sensorimotor training

SUMMARY:
Aging is associated with cognitive decline, ranging from normal to mild cognitive impairment or dementia. This leads to physical and cognitive impairment, which are risk factors for loss of autonomy therefore physical and cognitive training are important for cognitively impaired older adults. Cognitive somatosensory exercise (CSE) is a special comprehensive rehabilitation program for retraining sensory-induced motor control, and whole-body vibration (WBV), which enhances neuromuscular function, cognition, and balance. This study aims to investigate the effects of combined cognitive sensory-motor training with whole-body vibration on cognition and balance in older adults with mild to moderate cognitive impairment.

DETAILED DESCRIPTION:
A double-blinded randomized control trial will be conducted for ten months. The sample size was calculated through G-power and 50 participants will be recruited through the non-probability convenience sampling technique. Those who meet the inclusion criteria will be randomized into two groups (25 in the experimental group and 25 in the control group) through the online randomizer tool. The experimental group will receive cognitive sensorimotor training along with whole-body vibration. The control group will receive the cognitive sensorimotor training and Motor-cognitive dual-task training (mCdtt) simultaneously. Participants of each group will receive 60 minutes of training 3 times per week for 12 weeks. Outcome measures include the Montreal Cognitive Assessment (MoCA), the Stroop test will be used for the measurement of cognition and cognitive flexibility, the Mini bESTest for static and dynamic balance, and the Short physical performance battery for functional mobility. Assessment will be done at baseline, after the 6th week, 12th week, and at 16th week. Data analysis will be performed by using SPSS 26 software. Mixed ANOVA and repeated-measures ANOVA will be used for within-group analysis whereas between-group analysis will be performed by using one-way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Participants fulfilling given criteria will be included in this study

  * Both male and female participants will be included
  * The age limit for the participants will be 60 to 75
  * Participants with mild to moderate cognitive impairment having a Montreal Cognitive Assessment (MoCA) score of 13-25 (out of 30)
  * Participants with mild to moderate balance impairment having Mini BESTest cut-off score 13-28

Exclusion Criteria:

* Participants having given criteria will be excluded from this study

  * Participants having major depressive and anxiety disorder
  * Participants having significant visual and auditory impairment
  * Participants having a prior history of neurological disease or brain injury, and psychiatric disorders
  * Participants having cerebrovascular infarction
  * Participants having a neurological condition (epilepsy, loss of consciousness leading to a fall (e.g. vertigo syndrome)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA): | 12 weeks
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale with 12 subtasks in the MoCA test including memory, visuospatial orientation, executive functioning, phonemic fluency, two-item abstract thinking task, attention, concentration, working memory, language, and orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal. 18-25 points: Mild cognitive impairment. 10-17 points: Moderate cognitive impairment. Fewer than 10 points: Severe cognitive impairment. Inter-rater Reliability (0.96) Cronbach's alpha (0.79).
Mini Balance Evaluation Systems Test (Mini-BESTest): | 12 weeks
  The Mini-BESTest is a 14-item test that is a shortened version of the BESTest. It assesses important aspects of dynamic balance, including postural response to perturbation and gait stability. The Mini-BESTest has components of multiple individual balance assessments including items from the Berg Balance Scale, the Dynamic Gait Index, single-limb stance test, functional reach, Timed Up and Go, and modified Clinical Test of Sensory Interaction on Balance as well as a dual-task item and postural response items
Short physical performance battery (SPPB) | 12 weeks
  The Short Physical Performance Battery (SPPB) allows the evaluation of limitations in the functioning of the lower limbs concerning the lower limb strength by five chair lifts, the balance by the tandem/semi-tandem position, and the walking speed by the 4 m walk. Each component is scored from 0 to 4 and summed to yield scores between 0 (poor) and 12 (best) performance (31). The scores are added together to obtain an overall performance score, with a maximum of 12. A high score is defined as a score above 10, a medium score between 9 and 7, and a low score below 6. (32). Test-retest reliability of the SPPB was high: 0.87 (CI95%: 0.77-0.96)
The Stroop Color and Word Test (SCWT) | 12 weeks
  The Stroop test is a widely used executive function test to evaluate selective attention, speed of information processing, response inhibition and cognitive flexibility. In general, the Stroop effect occurs when individuals are presented with incongruent colour-word stimuli (e.g., the task requires to read the word "red" printed in blue ink or to name the colour of the ink instead of reading the word). Successful performance requires to inhibit an automatic behaviour (i.e., reading) in favour of a less practiced one (i.e., naming the colour of the ink). For all Stroop subtests, the completion times were the shortest for the individuals in the 18-29 age group with the highest education level and longest for the individuals in the 70-83 age group with the lowest education level. The test demonstrated acceptable internal consistency and high test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Society for the Rehabilitation of the Disabled (PSRD), Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No